CLINICAL TRIAL: NCT01895972
Title: A Single-Arm, Multicenter, Open-Label Study Evaluating the Long-Term Safety of Latanoprostene Bunod Ophthalmic Solution 0.024%, in Japanese Subjects With Open-Angle Glaucoma or Ocular Hypertension
Brief Title: Long-Term Safety of Latanoprostene Bunod Ophthalmic Solution 0.024% in Japanese Subjects With OAG or OHT
Acronym: JUPITER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 811
Record Dates: First submitted 2013-07-03; First posted 2013-07-11 (Estimated); Results first posted 2018-06-06 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-06

CONDITIONS: Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma; Ocular Hypertension | interventions — BOL 303259-X

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Latanoprostene Bunod (Experimental): Latanoprostene bunod 0.024% instilled into the eye once daily (QD) over a 1-year treatment period.
  Interventions: Drug: Latanoprostene bunod

INTERVENTIONS:
Drug: Latanoprostene bunod
  Other Names: BOL-303259-X

SUMMARY:
The objective of this study is to demonstrate the clinical safety of latanoprostene bunod 0.024% once daily (QD) over a 1-year treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a diagnosis of open angle glaucoma (OAG) (including normal-tension glaucoma [NTG],pigmentary or pseudoexfoliative glaucoma), or ocular hypertension (OHT) in one or both eyes.
* Subjects must meet the following IOP requirements at Visit 3 (Eligibility, Day 0[after washout for the subjects already on treatment]): mean/median IOP ≥15 mmHg and ≤36 mmHg at 10 AM in at least 1 eye; and IOP ≤36 mmHg in both eyes.
* Subjects with a corrected Decimal visual acuity (VA) or a Best-Corrected Decimal Visual Acuity (BCVA) of 0.5 or better in both eyes.

Exclusion Criteria:

* Subjects who are unable to discontinue contact lens use during and for 15 minutes following instillation of study drug and during study visits.
* Subjects who are unable to discontinue other eye drop medications such as artificial tears for 15 minutes prior to and 15 minutes after instillation of study drug.
* Subjects with a central corneal thickness greater than 600 μm in either eye.
* Subjects with any condition that prevents reliable applanation tonometry in either eye.
* Subjects with advanced glaucoma with a mean deviation (MD) < -12 dB, a history of split fixation, or a field loss threatening fixation in either eye.
* Subjects with any condition that prevents clear visualization of the fundus.
* Subjects who are monocular (fellow eye is absent).
* Subjects with aphakia in either eye.
* Subjects with an active corneal disease in either eye.
* Subjects with severe dry eye in either eye.
* Subjects with a history/diagnosis of a clinically significant or progressive retinal disease in either eye.
* Subjects with very narrow angles and subjects with angle closure congenital, or secondary glaucoma, and subjects with history of angle closure in either eye.
* Subjects with any intraocular infection or inflammation in either eye within 3 months prior to Visit 1 (Screening).
* Subjects with a history of ocular laser surgery in either eye within the 3 months (90 days) prior to Visit 1 (Screening).
* Subjects with a history of incisional ocular surgery or severe trauma in either eye within 3 months prior to Visit 1 (Screening).

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2013-07-05 (Actual); Primary Completion 2015-04-02 (Actual); Study Completion 2015-04-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason L. Vittitow, PhD, Study Director — Bausch & Lomb Incorporated
Locations (1):
- Bausch & Lomb Incorporated, Bridgewater, New Jersey, United States

REFERENCES:
- [Result] Kawase K, Vittitow JL, Weinreb RN, Araie M; JUPITER Study Group. Long-term Safety and Efficacy of Latanoprostene Bunod 0.024% in Japanese Subjects with Open-Angle Glaucoma or Ocular Hypertension: The JUPITER Study. Adv Ther. 2016 Sep;33(9):1612-27. doi: 10.1007/s12325-016-0385-7. Epub 2016 Jul 25. PMID 27457469

RESULTS

PARTICIPANT FLOW:
Groups:
- Latanoprostene Bunod: Latanoprostene bunod 0.024% instilled into the eye once daily (QD) over a 1-year treatment period.
  Latanoprostene bunod
Period: Overall Study
Arm/Group | Latanoprostene Bunod
Started | 130
Completed | 121
Not Completed | 9

BASELINE CHARACTERISTICS:
Arm/Group | Latanoprostene Bunod
Number analyzed (Participants) | 130
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.5 (10.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74
  Male | 56
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 130
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Japanese | 130
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 130

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Intraocular Pressure
Description: Change from baseline in intraocular pressure (IOP) following treatment with latanoprostene bunod 0.024% (instilled QD in the evening) with IOP assessed every 4 weeks from Week 4 to Week 52.
Time Frame: Baseline and week 4,8,12,16,20,24,28,32,36,40,44,48,52
Population: Safety population
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Latanoprostene Bunod
Number analyzed (Participants) | 130
mm Hg
  Week 4 | -4.30 (2.746)
  Week 8: number analyzed (Participants) | 129
  Week 8 | -4.57 (2.610)
  Week 12: number analyzed (Participants) | 128
  Week 12 | -4.76 (2.846)
  Week 16: number analyzed (Participants) | 126
  Week 16 | -4.79 (2.742)
  Week 20: number analyzed (Participants) | 126
  Week 20 | -4.94 (2.707)
  Week 24: number analyzed (Participants) | 126
  Week 24 | -4.94 (2.877)
  Week 28: number analyzed (Participants) | 126
  Week 28 | -4.93 (2.703)
  Week 32: number analyzed (Participants) | 125
  Week 32 | -5.04 (2.789)
  Week 36: number analyzed (Participants) | 123
  Week 36 | -5.32 (2.778)
  Week 40: number analyzed (Participants) | 122
  Week 40 | -5.25 (2.629)
  Week 44: number analyzed (Participants) | 122
  Week 44 | -5.12 (2.862)
  Week 48: number analyzed (Participants) | 122
  Week 48 | -5.12 (2.741)
  Week 52: number analyzed (Participants) | 121
  Week 52 | -5.25 (2.633)
Statistical Analysis 1: Comparison: Latanoprostene Bunod; comparison vs. baseline; Test type: Other; p < 0.001, t-test, 2 sided — The reduction from baseline in IOP was significant at all post-baseline assessment time points through Week 52

2. Primary Outcome: Clinical Safety
Description: Ocular adverse events reported over one year of once daily dosing of latanoprostene bunod 0.024%. Below is the percentage of subjects with >/=1 ocular AE Specifics of AEs are captured in the AE section.
Time Frame: 1 year
Population: Safety Population (Study Eye)
Measure: Count of Participants; unit: Participants
Arm/Group | Latanoprostene Bunod
Number analyzed (Participants) | 130
Participants | 76

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Latanoprostene Bunod
Serious Adverse Events (participants affected / at risk) | 5/130
Other Adverse Events (participants affected / at risk) | 76/130
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Latanoprostene Bunod (N=130)
Stomach cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
vestibular neuronitis (Infections and infestations) | 1
Car accident (Injury, poisoning and procedural complications) | 1
left tibia plateau fracture (Injury, poisoning and procedural complications) | 1
Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung ademocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Latanoprostene Bunod (N=130)
Abnormal sensation in the eye (Eye disorders) | 1
Asthenopia (Eye disorders) | 3
Blepheral pigmentation (Eye disorders) | 4
Blepharitis (Eye disorders) | 3
Cataract (Eye disorders) | 1
Conjunctival haemorrhage (Eye disorders) | 2
Conjunctival hyperemia (Eye disorders) | 23
Conjunctivitis allergic (Eye disorders) | 1
Conjunctivits bacterial (Eye disorders) | 1
Corneal erosion (Eye disorders) | 1
Dry eye (Eye disorders) | 1
Eczema eyelids (Eye disorders) | 1
Eye discharge (Eye disorders) | 1
Eye irritation (Eye disorders) | 15
Eye pain (Eye disorders) | 13
Eye pruritus (Eye disorders) | 3
Eyelid aedema (Eye disorders) | 1
Eyelid pruritus (Eye disorders) | 1
Foreign body in eye (Eye disorders) | 1
Foreign body sensation in eyes (Eye disorders) | 1
Growth of eyelashes (Eye disorders) | 21
Hordelolum (Eye disorders) | 1
Hypopigmentation of eyelid (Eye disorders) | 1
Iris hyperpigmentation (Eye disorders) | 5
Keratitis herpetic (Eye disorders) | 1
Ocular discomfort (Eye disorders) | 1
Punctate keratitis (Eye disorders) | 3
Trichiasis (Eye disorders) | 3
Visual impairment (Eye disorders) | 1
Vitreous floaters (Eye disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No